CLINICAL TRIAL: NCT04705168
Title: Performance of Nevisense Electrical Impedance Spectroscopy in Patients With Multiple Nevi and Large Acquired Nevi (LAN)
Brief Title: Study of the Nevisense Device to Assess Atypical Skin Lesions
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-010
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Nevus; Multiple Nevi; Large Acquired Nevi; Skin Lesion
Keywords: Atypical Skin Lesions; Skin Lesions; Multiple Nevi; Large Acquired Nevi; Memorial Sloan Kettering Cancer Center; 20-010
MeSH Terms: conditions — Nevus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants displaying nevi: Participants displaying a phenotype that consists of ≥ 100 nevi on the entire cutaneous surface and at least three large acquired nevi (LAN) > 5 mm in diameter. These patients have "atypical mole syndrome", which is a high-risk nevus phenotype and the target patient population in this study.
  Interventions: Diagnostic Test: Nevisense electrical impedance spectroscopy

INTERVENTIONS:
Diagnostic Test: Nevisense electrical impedance spectroscopy — Each participants will undergo Nevisense electrical impedance spectroscopy in order to characterize the electrical impedance spectroscopy scores of nevi in patients with ≥ 100 nevi on the entire cutaneous surface and at least three large acquired nevi (LAN) > 5 mm in diameter

SUMMARY:
The purpose of this study is to find out whether the Nevisense device can provide useful information about atypical moles to complement the usual assessments done during routine screening for melanoma. Assessing particpants' moles with the Nevisense device may help improve screening methods for the early detection of melanoma in people with atypical mole syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 30 years of age) at the time of the initial study visit.
* Patients displaying a phenotype that consists of ≥ 100 nevi on the entire cutaneous surface and at least three large acquired nevi (LAN) > 5 mm in diameter. These patients have "atypical mole syndrome", which is a high-risk nevus phenotype and the target patient population in this study.
* Patients with at least three clinically stable nevi between 5 and 20 mm in diameter.
* Patients (or LAR) who are able to provide informed consent.
* Patients with previous total body photography images taken at least 3 years prior

Exclusion Criteria:

* Patients without at least three clinically stable nevi between 5 and 20 mm in diameter.
* Patients with any electronic implantable devices.
* Patients who are pregnant (verbally confirmed with the participant).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan Kettering Cancer Center (MSKCC). If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. Potential subjects contacted by their treating physician will be referred to the investigator/research staff of the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Electrical impedance spectroscopy scores of participants' nevi | 2 weeks
  The primary objective is to characterize the electrical impedance spectroscopy scores of nevi in patients with ≥ 100 nevi on the entire cutaneous surface and at least three large acquired nevi (LAN) > 5 mm in diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq Marghoob, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org